CLINICAL TRIAL: NCT05547516
Title: A Prospective, Multicenter, Randomized Controlled Clinical Study of Blue Laser-5ALA-photodynamic Therapy (PDT) in the Prevention of Postoperative Tumor Recurrence in High-risk Non-muscle-invasive Bladder Cancer
Brief Title: Blue Laser -5ala Photodynamic Therapy (PDT) in High-Risk Non-muscle Invasive Bladder Cancer (NMIBC) Patients
Acronym: BL-PDT-RCT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2021ZDLSF02-16
Record Dates: First submitted 2022-09-14; First posted 2022-09-21 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: Non-muscle-invasive Bladder Cancer
MeSH Terms: conditions — Non-Muscle Invasive Bladder Neoplasms | interventions — Mitomycin; Epirubicin

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard infusion chemotherapy (including gemcitabine, mitomycin, Epirubicin, etc.) (Active Comparator): Standard infusion chemotherapy (including gemcitabine, mitomycin, epirubicin, etc.) was dissolved in 50mL normal saline or glucose and perfused into the bladder for 60min. Perfusion can be performed within 24 hours after surgery, and then once a week for a total of 8 times, and then once a month until 12 months after surgery.
  Interventions: Drug: Standard infusion chemotherapy
- BL-5ALA-PDT (Active Comparator): Bl-5ala-pdt protocol: 1.5g 5ALA, dissolved in 50mL normal saline, was infused into the bladder for 2h before surgery and before each cystoscopy, and blue laser irradiation was performed under flexible cystoscopy at 30mW/cm2 for 21min. PDT was performed during the operation and at 3, 6, and 9 months after the operation.
  Interventions: Drug: Standard infusion chemotherapy; Procedure: BL - 5 ala PDT

INTERVENTIONS:
Drug: Standard infusion chemotherapy — standard infusion chemotherapy (including gemcitabine, mitomycin, epirubicin, etc.), dissolved in 50mL normal saline or glucose, intravesical infusion chemotherapy, retained for 60min. Perfusion can be performed within 24 hours after surgery, and then once a week for a total of 8 times, and then once a month until 12 months after surgery
  Other Names: Standard infusion chemotherapy (including gemcitabine, mitomycin, Epirubicin, etc.)
Procedure: BL - 5 ala PDT — BL - 5 ala PDT - plan: 5ALA 1.5g (Shanghai Fudan-Zhangjiang Bio-Pharmaceutical Co.,Ltd), dissolved in 50mL normal saline, was infused into the bladder for 2 hours before surgery and before each cystoscopy. Blue laser irradiation was performed under a flexible cystoscope at 30mW/cm2 for 21min. PDT was performed during the operation and at 3, 6, and 9 months after the operation.
  Other Names: Blue laser-5ala Photodynamic therapy
  Arms: BL-5ALA-PDT

SUMMARY:
This project will conduct a large-sample, multi-center prospective clinical trial to further establish the safety and efficacy of BL-5ALA-PDT in preventing Non-Muscle Invasive Bladder Cancer (NMIBC) recurrence when compared to the usual postoperative perfusion chemotherapy regimen.

DETAILED DESCRIPTION:
This project will conduct a large-sample, multi-center prospective clinical trial to further establish the safety and efficacy of BL-5ALA-PDT in preventing Non-Muscle Invasive Bladder Cancer (NMIBC) recurrence when compared to the usual postoperative perfusion chemotherapy regimen.

Detailed Description:

1. Overall Study Design and Plan: a multicenter prospective randomized controlled clinical study;
2. Research steps: clinical recruitment, random enrollment, surgical treatment, regular postoperative preventive adjuvant intervention treatment + follow-up observation, and statistical analysis.
3. Screening Period: After obtaining the consent of the hospital ethics committee, the recruitment advertisement will be published to start the recruitment. September 1, 2022 to February 28, 2023, with at least one year follow-up. By reviewing inclusion and exclusion criteria, patients will be eligible to participate in the study. A total of 140 patients were recruited: 70 patients received conventional postoperative infusion chemotherapy (control group), and 70 patients received conventional postoperative infusion chemotherapy combined with BL-5ALA-PDT (BL-5ALA-PDT group).
4. Study Drug and PDT Administration: TURB-t uses the plasma resectoscope produced by Japan Olympus Company, and uses standardized layered electric resection or laser ablation surgical techniques; BL-5ALA-PDT uses Xi'an Lanji Medical Electronic Technology Co., Ltd. (The semiconductor laser therapeutic apparatus produced by Xi'an) was used as the PDT excitation light source, and 5ALA was purchased from Shanghai Fudan-zhangjiang Bio-Pharmaceutical Co., Ltd.
5. Postoperative infusion treatment plan: standard infusion chemotherapy (including gemcitabine, mitomycin, epirubicin, etc.), dissolved in 50 mL of normal saline or glucose, and intravesical infusion chemotherapy for 60 minutes. Perfusion can be done within 24 hours after operation, then once a week, a total of 8 times, and then changed to once a month to 12 months after operation; BL-5ALA-PDT program: 1.5g of 5ALA (Shanghai Fudan-zhangjiang Bio-Pharmaceutical Co., Ltd) was dissolved in 50 mL of normal saline, and infused into the bladder for 2 hours before surgery and before each cystoscopy. Blue laser irradiation was carried out at 30mW/cm2 and 21min under irradiation. PDT was performed during the operation and at 3, 6, and 9 months after the operation.
6. Postoperative follow-up plan: review urine routine, urinary B-ultrasound and cystoscopy in at 3, 6, and 9 months after operation, and record the follow-up in the follow-up registry at the same time. Follow-up content: urine routine, urinary B-ultrasound and cystoscopy results.
7. Evaluation indicators:

Main Outcome: Tumor recurrence rate 1 year after surgery Secondary Outcome: Observe postoperative complications (focus on side effects beyond standard perfusion therapy)

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically determined as high-risk NMIBC (meet any of the following: ①T1 stage tumor; ②G3 or high-grade urothelial carcinoma; ③CIS; cancer), patients planning to undergo transurethral surgery;
2. According to the EORTC score of 5 or above;
3. 18≤age≤80 years old, according to the requirements of the ethics committee, the patients (or authorized principals) agree to participate in this experiment and sign the informed consent.

Exclusion Criteria:

1. Patients with severe systemic diseases (such as severe coagulation disorders, decompensation of important organ functions) or chronic wasting diseases;
2. The patient has a history of other malignant tumors in the past five years;
3. Pregnant and lactating women;
4. Those who have undergone major surgery within 1 month before enrollment;
5. Participate in other clinical trials;
6. Other conditions (such as: mental illness, etc.) considered inappropriate by the researcher.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2022-09-13 (Estimated); Primary Completion 2022-09-13 (Estimated); Study Completion 2024-02-01 (Estimated)

PRIMARY OUTCOMES:
Tumor recurrence rate 1 year after surgery | from date of randomization until the date of first documented Tumor recurrence
  The recurrence rate of NMBC at 1 year after surgery was evaluated by regular urine routine, urinary B-ultrasound and cystoscopy

SECONDARY OUTCOMES:
Observe postoperative complications (focus on side effects beyond standard perfusion therapy) | from date of randomization until the date of first documented postoperative complications
  postoperative complications were evaluated by regular urine routine, urinary B-ultrasound and cystoscopy

CONTACTS AND LOCATIONS:
Overall Officials: Dalin He, Dr., Principal Investigator — First Affiliated Hospital Xi'an Jiaotong University
Locations (1):
- Dalin He, Xi'an, Shaanxi, China

REFERENCES:
- [Background] Babjuk M, Burger M, Comperat EM, Gontero P, Mostafid AH, Palou J, van Rhijn BWG, Roupret M, Shariat SF, Sylvester R, Zigeuner R, Capoun O, Cohen D, Escrig JLD, Hernandez V, Peyronnet B, Seisen T, Soukup V. European Association of Urology Guidelines on Non-muscle-invasive Bladder Cancer (TaT1 and Carcinoma In Situ) - 2019 Update. Eur Urol. 2019 Nov;76(5):639-657. doi: 10.1016/j.eururo.2019.08.016. Epub 2019 Aug 20. PMID 31443960
- [Background] Messing EM, Tangen CM, Lerner SP, Sahasrabudhe DM, Koppie TM, Wood DP Jr, Mack PC, Svatek RS, Evans CP, Hafez KS, Culkin DJ, Brand TC, Karsh LI, Holzbeierlein JM, Wilson SS, Wu G, Plets M, Vogelzang NJ, Thompson IM Jr. Effect of Intravesical Instillation of Gemcitabine vs Saline Immediately Following Resection of Suspected Low-Grade Non-Muscle-Invasive Bladder Cancer on Tumor Recurrence: SWOG S0337 Randomized Clinical Trial. JAMA. 2018 May 8;319(18):1880-1888. doi: 10.1001/jama.2018.4657. PMID 29801011
- [Background] Agostinis P, Berg K, Cengel KA, Foster TH, Girotti AW, Gollnick SO, Hahn SM, Hamblin MR, Juzeniene A, Kessel D, Korbelik M, Moan J, Mroz P, Nowis D, Piette J, Wilson BC, Golab J. Photodynamic therapy of cancer: an update. CA Cancer J Clin. 2011 Jul-Aug;61(4):250-81. doi: 10.3322/caac.20114. Epub 2011 May 26. PMID 21617154
- [Background] Railkar R, Agarwal PK. Photodynamic Therapy in the Treatment of Bladder Cancer: Past Challenges and Current Innovations. Eur Urol Focus. 2018 Jul;4(4):509-511. doi: 10.1016/j.euf.2018.08.005. Epub 2018 Aug 23. PMID 30145112
- [Background] Kushibiki T, Hirasawa T, Okawa S, Ishihara M. Blue laser irradiation generates intracellular reactive oxygen species in various types of cells. Photomed Laser Surg. 2013 Mar;31(3):95-104. doi: 10.1089/pho.2012.3361. Epub 2013 Feb 7. PMID 23390956
- [Background] Ericson MB, Grapengiesser S, Gudmundson F, Wennberg AM, Larko O, Moan J, Rosen A. A spectroscopic study of the photobleaching of protoporphyrin IX in solution. Lasers Med Sci. 2003;18(1):56-62. doi: 10.1007/s10103-002-0254-2. PMID 12627275